CLINICAL TRIAL: NCT02716792
Title: Randomized, Open Label Study to Evaluate Renal Safety of Intravenous Bondronat 6 mg Infusions Over 15 Minutes Versus 60 Minutes in Patients With Metastatic Bone Disease Due to Breast Cancer
Brief Title: A Study to Evaluate Renal Safety of Intravenous Ibandronate (Bondronat) in Participants With Metastatic Bone Disease Due to Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19188
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Bone Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid

ARMS (2):
- Ibandronate 15-Minute Infusion (Experimental): Participants will receive ibandronate IV infusions over a 15-minute interval.
  Interventions: Drug: Ibandronate
- Ibandronate 60-Minute Infusion (Active Comparator): Participants will receive ibandronate IV infusions over a 60-minute interval.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Participants will receive ibandronate, 6 mg via IV infusion, every 3 weeks for up to 9 cycles. The infusion interval will be either 15 or 60 minutes depending upon treatment group assignment every 3 weeks (9 treatment cycles in total).
  Other Names: Bondronat

SUMMARY:
This study will evaluate renal function in participants with metastatic bone disease due to breast cancer receiving intravenous (IV) infusions of ibandronate (Bondronat) 6 milligrams (mg), over either 15 minutes or 60 minutes, every 3 weeks. Efficacy and safety of ibandronate in the 2 groups of participants will also be compared. The anticipated time on study treatment is 7 months, and the target sample size is 318 individuals.

ELIGIBILITY:
Inclusion Criteria:

* For participants of childbearing potential: negative pregnancy test and ready to use effective contraceptive measures
* Metastatic breast cancer with at least one bone metastasis
* Karnofsky index >/= 60
* Life expectancy >/= 6 months
* Estimated creatinine clearance (Cockcroft and Gault formula) >/= 30 milliliters per minute (mL/min)

Exclusion Criteria:

* Pregnancy or breast feeding participant
* Participant who had a current dental problem, particularly tooth or jaw infection, trauma or surgery on tooth or jaw in the previous six weeks, medical history of jaw osteonecrosis or delayed healing after dental surgery
* Participant who was participating or had participated in the last 30 days to a clinical trial investigating treatments
* Uncontrolled brain metastasis
* Severe or concomitant infection
* Known medical history of systemic disease with renal lesion
* Rapidly progressing renal failure at inclusion
* Uncontrolled cardiac disorder
* Hypercalcaemia (> 2.7 millimoles per liter [mmol/L]), hypocalcaemia (< 2 mmol/L)
* Participant receiving nephrotoxic chemotherapy
* Participant eligible for haematopoietic stem cell transplantation at inclusion time
* Bisphosphonate therapy in the 3 weeks before randomization
* Known hypersensitivity to ibandronate or other bisphosphonates

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Creatinine clearance (CrCl) Estimated by Cockcroft-Gault Formula | 28 days after last infusion (approximately 2 years)

SECONDARY OUTCOMES:
Number of Participants with Bone Pain According to Visual Analog Scale (VAS) | Every 3 weeks up to approximately 6 months
Number of Participants With of Skeletal Events (Vertebral and Non-Vertebral Fractures, Impending Fracture, Radiotherapy or Surgery to Bone) | Up to approximately 7 months
Percentage of Participants on Analgesics According to World Health Organization (WHO) Three-Step Analgesic Ladder | Up to approximately 7 months
Karnofsky Index score | Every 3 weeks up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (28):
- France (28):
  - Amboise
  - Angers
  - Bayonne
  - Besançon
  - Boulogne-Billancourt
  - Brest
  - Chambéry
  - Clermont-Ferrand
  - Évreux
  - Gap
  - Hyères
  - Le Chesnay
  - Metz-Tessy
  - Nantes
  - Neuilly-sur-Seine
  - Paris
  - Rennes
  - Rouen
  - Saint-Brieuc
  - Saint-Cloud
  - Saint-Grégoire
  - Saint-Jean
  - Salouël
  - Strasbourg
  - Trappes
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Villejuif